CLINICAL TRIAL: NCT06458010
Title: Clinical Exploration Trial of YOLT-101 in the Treatment of Familial Hypercholesterolemia (FH)
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FH-YOLT-101-001
Record Dates: First submitted 2024-05-17; First posted 2024-06-13 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Familial Hypercholesterolemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II

STUDY DESIGN:
Intervention Model Description: 0.2mg/kg, 0.4mg/kg, 0.6mg/kg, 40mg, 50mg
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single Arm (Experimental): dosage group: 0.2mg/kg, 0.4mg/kg, 0.6mg/kg,40mg,50mg; dosage form: injection; frequency of administration: once.
  Interventions: Drug: YOLT-101

INTERVENTIONS:
Drug: YOLT-101 — The IP is administered intravenously at the predetermined dose.

SUMMARY:
This study is a single arm, open, single dose escalation trial aimed at evaluating the safety and tolerability of YOLT-101 administration in patients with familial hypercholesterolemia; Determination of YOLT-101 OBD; Preliminary evaluation of the effects of single administration of YOLT-101 on plasma lipid and lipoprotein levels.

Note: OBD is defined as the dosage at which plasma PCSK9 protein levels decrease between 60% and 95% from baseline on the 28th day after YOLT-101 administration. OBD ≤ Maximum Tolerable Dose (MTD).

In this study, the longest screening period for the main study was 42 days, the treatment day was Day 1 (D1), and the safe follow-up period was up to 52 weeks after medication. In the main study, when OBD occurs, additional subjects will be added to the dose group (specific number of cases will be negotiated between the cooperating organization and investigators) for further validation. In addition, subjects in the first dose group can voluntarily receive a second drug administration of OBD level.

After the completion of the main study, participants will undergo long-term follow-up. According to the Technical Guidelines for Long term Follow up Clinical Research of Gene Therapy Products (Trial) released by CDE, a long-term follow-up until 15 years after the medicine administration is required .

DETAILED DESCRIPTION:
Protocol (V1.2, 6 May 2024) has been approved on 14 May 2024 Protocol (V1.3 ,23 May 2024) has been approved on 12 Jun 2024 Protocol (V1.4 ,24 Jun 2024) has been approved on 15 Jul 2024 Protocol (V1.5 ,18 Oct 2024) has been approved on 28 Oct 2024 Protocol (V1.6 ,27 Nov 2024) has been approved on 27 Dec 2024 Protocol (V1.7 ,6 Jan 2025) has been approved on 27 Jan 2025 Protocol (V1.8 ,19 Feb 2025) has been approved on 24 Mar 2025

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged 18 to 75 years inclusive, at the time of signing informed consent.
2. Meets the diagnostic criteria for familial hypercholesterolemia.
3. At screening, there is a mutation in the PCSK9 and/or ApoB and/or LDLR gene.
4. At screening, weight is ≥40kg, and Body Mass Index (BMI) is >18kg/m^2.
5. At screening, subjects must meet the following laboratory criteria:

   5.1 Hematology: Absolute Neutrophil Count (ANC) ≥1.5×10^9/L, Platelet (PLT) ≥100×10^9/L, Hemoglobin (HGB) ≥90 g/dL; 5.2 Liver Function: Aspartate Aminotransferase (AST), Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP) <2.0×Upper Limit of Normal (ULN), Total Bilirubin (TBIL) ≤1.5×ULN; 5.3 Renal Function: Serum Creatinine (Cr) ≤1.5×ULN, and Glomerular Filtration Rate (GFR) >60mL/min*1.73m^2; 5.4 Coagulation Function: Prothrombin Time (PT), Activated Partial Thromboplastin Time (APTT), International Normalized Ratio (INR) <1.5×ULN; 5.5 Fasting Triglycerides <5.6mmol/L.
6. On moderate intensity or higher statin therapy (statin treatment stable for 4 weeks) with LDL-C ≥2.6mmol/L; for those with evidence of atherosclerosis, LDL-C ≥1.8mmol/L. (Evidence of atherosclerosis includes: 1. History of myocardial infarction, angina, coronary artery revascularization, non-embolic ischemic stroke or transient ischemic attack, intermittent claudication; 2. Presence of advanced subclinical atherosclerosis: Coronary artery calcium score > 100 Agatston units, or above the 75th percentile for age and sex; or coronary artery CT angiography showing stenosis > 50%, or multiple vessels with non-obstructive plaques.)
7. Subjects and their partners must use effective contraceptive measures during the study period and for at least 6 months after the end of the main study.
8. Voluntarily sign informed consent.

Exclusion Criteria:

1. Within at least 14 days (or 5 half-lives of the drug, whichever is longer, for small molecule/small nucleic acid drugs) or 2 months (for biological agents such as PCSK9 inhibitors) or 1 year (for PCSK9 small nucleic acid drugs) before accepting the study medication, those who have used prescription drugs that affect lipid metabolism other than statins, or those who have used any non-prescription drugs affecting lipid metabolism within at least 14 days before accepting the study medication (such as traditional Chinese medicine/patent Chinese medicine, vitamins, fish oil (>1000mg/day), drugs or health products containing red yeast rice, etc.; except for those who have been on stable non-cyclic hormone replacement therapy for more than 8 weeks and agree not to change the treatment plan for at least 28 days after receiving the trial medication); those who are currently participating in other clinical studies of lipid-lowering drugs and have used study medication.
2. Patients with poorly controlled hypertension (systolic blood pressure (SBP) ≥160mmHg and/or diastolic blood pressure (DBP) ≥100mmHg).
3. Patients with poorly controlled diabetes (glycated hemoglobin >8.5%).
4. Those allergic to drugs or components of LNP-mRNA vaccines contained in lipid nanoparticles (LNP), or those who have experienced adverse reactions due to LNP-based drug treatment, such as: 4.1 After receiving LNP-based drug treatment, ALT or AST > 3.0×ULN; 4.2 After receiving LNP-based drug treatment, INR > 1.5 or APTT/d-dimer > 1.5×ULN; 4.3 Any infusion reaction that requires clinical intervention or slows down or stops the infusion of LNP-based drug treatment; 4.4 Any other adverse reactions deemed related to LNP-based drug treatment by the investigator.
5. Within 3 months before screening, those who smoke more than 5 cigarettes per day or consume an equivalent amount of nicotine or nicotine replacement products.
6. Within 3 months before screening, those with a history of alcohol abuse [consuming more than 14 units of alcohol per week (1 unit ≈ 360mL beer or 45mL of liquor with 40% alcohol or 150mL of wine)]; or those who test positive for alcohol breath research at screening or admission.
7. At screening, those with New York Heart Association (NYHA) defined class III-IV heart failure, or left ventricular ejection fraction <50%, or prolonged QTc interval (females >470ms, males >450ms).
8. Within 3 months before screening, those with poorly controlled severe arrhythmias, such as recurrent and highly symptomatic ventricular tachycardia, rapid ventricular response atrial fibrillation, or supraventricular tachycardia that is not well controlled with medication.
9. Within 3 months before screening, those with myocardial infarction, unstable angina, percutaneous coronary intervention, coronary artery bypass grafting, severe deep vein thrombosis, or pulmonary embolism; those who have had a cerebrovascular accident within 6 months before screening or plan to undergo cardiac surgery or revascularization during the main study period.
10. Those with diseases that significantly affect lipid levels and are uncontrollable, such as nephrotic syndrome, severe liver disease, Cushing's syndrome, thyroid dysfunction, etc. (those with hypothyroidism before screening who have been on stable thyroid replacement therapy for ≥28 days, with normal TSH testing, and agree to maintain the thyroid replacement drug dose unchanged during the study may be considered for inclusion).
11. Those who have donated more than 500 mL of blood within 3 months before screening.
12. Those who cannot or are unwilling to accept the required medication treatment plan before treatment.
13. Those who have undergone antithrombotic treatment (such as warfarin, dabigatran, apixaban) within 14 days before enrollment.
14. Those with a history of easy bleeding or coagulation disorders (such as liver cirrhosis, malignant hematological diseases, antiphospholipid antibody syndrome).
15. Those with an expected survival of less than 2 years.
16. Those known or suspected to have systemic viral, parasitic, or fungal infections, or those expected to receive antibiotic treatment within 14 days after screening.
17. Those who test positive for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody at screening.
18. Those who have undergone liver, heart, or other solid organ transplantation or bone marrow transplantation within 1 year before screening or plan to undergo transplantation during the trial period.
19. Those with a history of malignant tumors within 5 years before screening (except for cured basal cell carcinoma of the skin, squamous cell carcinoma of the skin, cervical carcinoma in situ, low-grade prostatic intraepithelial neoplasia, and cured basal cell carcinoma of the thyroid).
20. Those with a history of drug abuse within 3 years before screening.
21. Women who are pregnant or breastfeeding.
22. Those with other hematopoietic system, digestive system, or central nervous system (including cerebrovascular diseases, degenerative diseases) diseases that the investigator believes will interfere with evaluation or limit participation in the trial.
23. Those with severe mental illnesses that the investigator believes cannot be adequately controlled by drug treatment.
24. Those unwilling to comply with the research procedures or unwilling to fully cooperate.
25. Other situations deemed by the investigator as not suitable for participation in clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
safety evaluation of YOLT-101 | through week 52
  The safety of YOLT-101 evaluated by the proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs).

SECONDARY OUTCOMES:
pharmacokinetics of YOLT-101 | through Day 28
  The Peak Plasma Concentration (Cmax) of YOLT-101. 0.5 predose,2,12,24,48,72,144,312,648hours.
pharmacodynamics | through week 52
  The effect of YOLT-101 on serum levels of LDL-C
pharmacodynamics | through week 52
  The effect of YOLT-101 on plasma levels of PCSK9
pharmacokinetics of YOLT-101 | through Day 28
  Area under the plasma concentration versus time curve (AUC); 0.5 predose,2,12,24,48,72,144,312,648hours.
pharmacokinetics of YOLT-101 | through Day 28
  Tmax;
pharmacokinetics of YOLT-101 | through Day 28
  T1/2

CONTACTS AND LOCATIONS:
Locations (1):
- Deparment of Liver Surgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No